CLINICAL TRIAL: NCT00108875
Title: Vaccination of Patients With Advanced Melanoma, Pancreatic, Colon and Cervical Cancer With HLA-A1, -A2 and -B35 Restricted Survivin Peptides
Brief Title: Survivin Peptide Vaccination for Patients With Advanced Melanoma, Pancreatic, Colon and Cervical Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Julius-Maximilians University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SuMo-Sec-01; PEI 0899/01; IRB 07/03
Record Dates: First submitted 2005-04-19; First posted 2005-04-20 (Estimated); Last update posted 2006-07-28 (Estimated); Status verified 2005-06

CONDITIONS: Malignant Melanoma; Pancreatic Cancer; Colon Cancer; Cervical Cancer
Keywords: Peptide vaccine therapy; Survivin
MeSH Terms: conditions — Melanoma; Pancreatic Neoplasms; Colonic Neoplasms; Uterine Cervical Neoplasms

INTERVENTIONS:
Biological: Survivin peptide vaccine

SUMMARY:
This study evaluates the safety, the immunological response and the clinical outcome of a vaccination with survivin peptides for patients with advanced melanoma, pancreatic, colon and cervical carcinoma.

DETAILED DESCRIPTION:
As prognosis of advanced melanoma, pancreatic, colon and cervical cancer remains gloomy, new therapeutic modalities have to be developed to improve the patient´s clinical outcome. Immunotherapy, which targets tumor associated antigens of tumor cells or tumor stroma, is currently an intensively investigated, novel therapeutic option. As survivin is expressed both by neoplastic cells as well as by endothelial cells of the tumor vasculature, this antigen is an intriguing target molecule. Spontaneous cytotoxic T-cell responses against different survivin epitopes in cancer patients underline the relevance of survivin-directed immunological trials. This study is comprised of a peptide vaccine with HLA-A1, -A2 and -B35 restricted survivin epitopes in Montanide ISA-51 for patients with stage IV melanoma, advanced pancreatic, colon and cervical carcinoma. The vaccine is applicated as a deep subcutaneous injection. Vaccination is administered for the first 2 months weekly, afterwards every 4 weeks. Standard staging examinations are performed every three months. Clinical, laboratory and immunological monitoring is done every month.Diagnostic leucapheresis is performed before first vaccination and afterwards every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Advanced melanoma, pancreatic, colon and cervical cancer
* At least 1 prior postoperative conventional therapy (chemotherapy, radiation, immunotherapy)
* HLA-A1, -A2, -B35
* More than 4 weeks since last chemo-, immune- or radiotherapy
* ECOG-PS (Eastern Cooperative Oncology Group- Performance Status) of 0-1
* Sufficient renal, hepatic and bone marrow function: thrombocytes > 75.000/ul; hb > 9 g/dl; leucocytes > 2.500/ul; creatinine < 2 mg/dl; GOT/GPT < twice the normal value
* negative for HIV and Hbs
* Older than 18 years
* Informed consent

Exclusion Criteria:

* Acute/chronic infections
* Positive for HIV, Hbs
* Autoimmune disorders
* Pregnancy, breast feeding

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2003-04

PRIMARY OUTCOMES:
Progression-free survival
Overall survival
Immunological response

SECONDARY OUTCOMES:
Best response

CONTACTS AND LOCATIONS:
Overall Officials: Juergen C Becker, MD, Principal Investigator — Department of Dermatology, University of Wuerzburg, Germany
Locations (1):
- Julius-Maximilians-University of Wuerzburg, Germany, Department of Dermatology, Würzburg, Bavaria, Germany

REFERENCES:
- [Background] Blanc-Brude OP, Mesri M, Wall NR, Plescia J, Dohi T, Altieri DC. Therapeutic targeting of the survivin pathway in cancer: initiation of mitochondrial apoptosis and suppression of tumor-associated angiogenesis. Clin Cancer Res. 2003 Jul;9(7):2683-92. PMID 12855648
- [Background] Otto K, Andersen MH, Eggert A, Keikavoussi P, Pedersen LO, Rath JC, Bock M, Brocker EB, Straten PT, Kampgen E, Becker JC. Lack of toxicity of therapy-induced T cell responses against the universal tumour antigen survivin. Vaccine. 2005 Jan 4;23(7):884-9. doi: 10.1016/j.vaccine.2004.08.007. PMID 15603888
- [Background] Andersen MH, Pedersen LO, Capeller B, Brocker EB, Becker JC, thor Straten P. Spontaneous cytotoxic T-cell responses against survivin-derived MHC class I-restricted T-cell epitopes in situ as well as ex vivo in cancer patients. Cancer Res. 2001 Aug 15;61(16):5964-8. PMID 11507035
- [Background] Andersen MH, Pedersen LO, Becker JC, Straten PT. Identification of a cytotoxic T lymphocyte response to the apoptosis inhibitor protein survivin in cancer patients. Cancer Res. 2001 Feb 1;61(3):869-72. PMID 11221872
- [Background] Kim HS, Shiraki K, Park SH. Expression of survivin in CIN and invasive squamous cell carcinoma of uterine cervix. Anticancer Res. 2002 Mar-Apr;22(2A):805-8. PMID 12014654
- [Background] Reker S, Becker JC, Svane IM, Ralfkiaer E, Straten PT, Andersen MH. HLA-B35-restricted immune responses against survivin in cancer patients. Int J Cancer. 2004 Mar 1;108(6):937-41. doi: 10.1002/ijc.11634. PMID 14712500
- [Background] Reker S, Meier A, Holten-Andersen L, Svane IM, Becker JC, thor Straten P, Andersen MH. Identification of novel survivin-derived CTL epitopes. Cancer Biol Ther. 2004 Feb;3(2):173-9. doi: 10.4161/cbt.3.2.611. Epub 2004 Feb 1. PMID 14726703